CLINICAL TRIAL: NCT05566314
Title: Amunizer for Immune Support: A Randomized, Placebo Controlled, Double Blind Clinical Trial
Brief Title: Beverage for Immune Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Principal Investigator, Jessie Hawkins, President, Nutraceuticals Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-06-3600
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Immune

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Herbal and probiotic beverage
  Interventions: Dietary Supplement: Amunizer
- Placebo (Placebo Comparator): Similar beverage without the probiotics and botanicals
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Amunizer — 12 oz. herbal, probiotic and antioxidant herbal beverage
  Arms: Intervention
Other: Placebo — 12 oz. flavored beverage
  Arms: Placebo

SUMMARY:
Evaluate the effects of a beverage supplement on immune health over an 8 week intervention using either a placebo or active supplement.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of days with symptoms documented by the Franklin Health Immune Inventory (FHII) | from baseline to the end of the study, 8 weeks
  The FHII measures incidence and severity of over 50 signs of immune health. Days with symptoms will range from 0 to 56 days, indicating no sickness to sick every day.
Severity of symptoms documented by the FHII | from baseline to the end of the study, 8 weeks
  The FHII measures incidence and severity of over 50 signs of immune health. Symptom severity is measured on a likert scale with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Incidence and severity on the upper respiratory symptom subscale of the FHII | from baseline to the end of the study, 8 weeks
  The FHII subscale measures 16 respiratory symptoms on a likert scale with higher scores indicating greater severity.
Incidence and severity on the gastrointestinal symptom subscale of the FHII | from baseline to the end of the study, 8 weeks
  The FHII subscale measures 11 gastrointestinal symptoms on a likert scale with higher scores indicating greater severity.
Incidence and severity on the dermal symptom subscale of the FHII | from baseline to the end of the study, 8 weeks
  The FHII subscale measures 9 dermal symptoms on a likert scale with higher scores indicating greater severity.
Change from baseline scores on the Franklin Energy Level Inventory | 8 week
  The Franklin Energy Level Inventory measures signs of energy across 6 subdomains, with higher scores indicating greater levels of energy.
Change from baseline scores on the Franklin Sleep Quality Inventory | 8 week
  The Franklin Sleep Quality Inventory measures sleep quality across 7 subdomains, with higher scores indicating higher quality sleep.
Change from baseline scores on the Franklin Mood Scale | 8 week
  The Franklin Mood Scale measures mood stats across 4 subdomains, with higher scores indicating improvements to mood.

CONTACTS AND LOCATIONS:
Locations (1):
- Franklin Health Research Center, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No